CLINICAL TRIAL: NCT04653129
Title: Use of Autologous Fat to Improve Functional Outcomes After Upper Limb Nerve Injuries
Brief Title: Autologous Fat in Peripheral Nerve Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed ElSayed Sharaf Ahmed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fat for Nerve Injury
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Nerve Injury
Keywords: fat graft; autologous fat; peripheral nerve injury
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the assessment of outcome measures will be performed by a dedicated surgeon not involved in the surgery or preoperative patient evaluation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): Primary nerve repair with autologous fat graft (Experimental): Standard nerve repair will be performed with 9/0 nylon sutures, under magnification by an operating microscope with autologous fat grafting around site of repair
  Interventions: Procedure: Autologous Fat Grafting; Procedure: Primary Nerve Repair
- Group (B): Standard primary nerve repair (Active Comparator): Standard nerve repair will be performed with 9/0 nylon sutures, under magnification by an operating microscope without fat grafting.
  Interventions: Procedure: Primary Nerve Repair

INTERVENTIONS:
Procedure: Autologous Fat Grafting — * The fat grafts will be harvested from the abdomen or lateral thighs in a closed sterile system, then prepared according to Coleman guidelines. The blood and oil layers are then separated from the adipose tissue.
  * The lipoaspirate will be injected based on a technique described by Vaienti et al, by 17-gaug cannula which will be inserted through the skin around the main incision at the nerve repair site, and the fat graft will be injected after closure of the skin.
  Arms: Group (A): Primary nerve repair with autologous fat graft
Procedure: Primary Nerve Repair — Standard Epineural nerve repairs will be performed with 9/0 nylon sutures, under magnification by an operating microscope.

SUMMARY:
The aim of this study is to assess the efficacy of autologous fat graft in enhancing peripheral nerve regeneration. The investigators hypothesize that fat grafting will allow for faster and greater recovery of motor and sensory function following surgical repair of injured peripheral nerves.

DETAILED DESCRIPTION:
Traumatic injuries to peripheral nerves are a frequent finding after hand trauma. High morbidity after nerve injuries mainly affects the younger and working population, with consequent decrease in life quality and productivity .

Even in direct nerve repair and microsurgical nerve coaptation, regeneration is often suboptimal with incomplete target reinnervation. Suboptimal outcome is attributed to axonal degeneration, fibrotic scar formation, and neuromas at the site of injury.

The use of adipose tissue has become very popular in tissue engineering and reconstructive surgery in recent years. It is proposed as a "regenerative tool" for various tissues, including peripheral nerves, because it offers an effective and minimally invasive procedure for obtaining stem cells.

Unprocessed fat grafting can provide a simple approach to improve peripheral nerve regeneration by means of neoangiogenesis & inflammatory response modulation. Furthermore, it serves as a good protective barrier in peripheral nerve surgery, reducing fibrosis and adhesions.

A recent study advocated by Tuncel et al, concluded that combined use of autologous fat graft with surgical repair methods induced significantly better regeneration in rats [3]. In another study by Kilic et al, using adipose tissue flap in a crush injury model in rats was found to be superior to other groups in myelin thickness, nerve fiber density, axon count, and functional recovery at 4 weeks. They concluded that fat tissue seems to promote nerve regeneration because of its stem cell content.

To our knowledge, no prior studies have examined the use of fat graft in peripheral nerve repair in humans. So, the investigators proposed this clinical study to evaluate the outcomes of primary nerve repair combined with autologous fat graft in peripheral nerve injuries.

ELIGIBILITY:
Inclusion Criteria:

- Acute median or ulnar nerve lacerations below elbow

Exclusion Criteria:

* Old Nerve lacerations > 48 hours
* Nerve gap which requires nerve grafting
* Psychosocial issues that would limit participation and compliance

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Modified British Medical Research Council, sensory grading | 6-12 months
  standardized clinical assessment of sensory function using two-point discrimination and monofilament testing by a score from S0 to S4; the higher score indicates better sensation
Modified British Medical Research Council, motor grading | 6-12 months
  standardized clinical assessment of motor function on a scale from M0 to M5; the higher score indicates better strength.

SECONDARY OUTCOMES:
Nerve conduction study | 6-12 months
  measure for amplitude of response, latency of response and velocity of response measurements.
Disability of the Arm, Shoulder, and Hand (DASH) score | 6-12 months
  self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100 (most severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek A El-Gammal, MD, Study Director — Assiut University Hospital - Orthopaedics & Traumatology Dept.; Youssef S Hassan, MD, Study Chair — Assiut University Hospitals - Plastic Surgery Dept.; Awny M Asklany, MD, Study Director — Assiut University Hospitals - Plastic Surgery Dept.; Ahmed S Sharaf, MsC, Principal Investigator — Assiut University Hospitals - Plastic Surgery Dept.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Summa PG, Schiraldi L, Cherubino M, Oranges CM, Kalbermatten DF, Raffoul W, Madduri S. Adipose Derived Stem Cells Reduce Fibrosis and Promote Nerve Regeneration in Rats. Anat Rec (Hoboken). 2018 Oct;301(10):1714-1721. doi: 10.1002/ar.23841. Epub 2018 Jul 10. PMID 29710394
- [Background] Ngeow WC. Scar less: a review of methods of scar reduction at sites of peripheral nerve repair. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Mar;109(3):357-66. doi: 10.1016/j.tripleo.2009.06.030. PMID 20219599
- [Background] Tuncel U, Kostakoglu N, Turan A, Cevik B, Cayli S, Demir O, Elmas C. The Effect of Autologous Fat Graft with Different Surgical Repair Methods on Nerve Regeneration in a Rat Sciatic Nerve Defect Model. Plast Reconstr Surg. 2015 Dec;136(6):1181-1191. doi: 10.1097/PRS.0000000000001822. PMID 26273733
- [Background] Walocko FM, Khouri RK Jr, Urbanchek MG, Levi B, Cederna PS. The potential roles for adipose tissue in peripheral nerve regeneration. Microsurgery. 2016 Jan;36(1):81-8. doi: 10.1002/micr.22480. Epub 2015 Sep 7. PMID 26773850
- [Background] Kilic A, Ojo B, Rajfer RA, Konopka G, Hagg D, Jang E, Akelina Y, Mao JJ, Rosenwasser MP, Tang P. Effect of white adipose tissue flap and insulin-like growth factor-1 on nerve regeneration in rats. Microsurgery. 2013 Jul;33(5):367-75. doi: 10.1002/micr.22101. Epub 2013 May 7. PMID 23653396
- [Background] Iannace C, Di Libero L, Manetta F, Sciascia V, Pizza A, Napolitano S, Ferraro A, Scetta G, Esposito D, Varriale S, Candela G, Caracciolo F. [Coleman lipofilling: experience of an Italian group and review of the literature]. Chir Ital. 2009 Jan-Feb;61(1):67-75. Italian. PMID 19391342
- [Background] Vaienti L, Gazzola R, Villani F, Parodi PC. Perineural fat grafting in the treatment of painful neuromas. Tech Hand Up Extrem Surg. 2012 Mar;16(1):52-5. doi: 10.1097/BTH.0b013e31823cd218. PMID 22411121